CLINICAL TRIAL: NCT03540329
Title: Comparative Study Between Internal and External Distraction Osteogenesis in Lower Face Asymmetry
Brief Title: Comparison Between Internal and External Distractors in Osteogenesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ehab Ragab, Assistant Lecturer, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Distraction osteogenesis
Record Dates: First submitted 2018-03-25; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Micrognathia of Lower Jaw; Retrognathism; Facial Asymmetry
Keywords: osteogenesis; distraction; Lower face asymmetry
MeSH Terms: conditions — Micrognathism; Retrognathia; Facial Asymmetry

STUDY DESIGN:
Intervention Model Description: Cohort prospective study model comparing two different techniques for distraction osteogenesis in 4 different subgroups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- I-A Internal distraction (Active Comparator): Internal osteogenesis distractor in congenital mandibular deformities in patients in growing age.
  Interventions: Device: Internal Osteogenesis distractor
- I-A External distraction (Active Comparator): External osteogenesis distractor in congenital mandibular deformities in patients in growing age.
  Interventions: Device: External Osteogenesis distractor
- I-B Internal distraction (Active Comparator): Internal osteogenesis distractor in congenital mandibular deformities in adult patients.
  Interventions: Device: Internal Osteogenesis distractor
- I-B External distraction (Active Comparator): External osteogenesis distractor in congenital mandibular deformities in adult patients.
  Interventions: Device: External Osteogenesis distractor
- II-A Internal distraction (Active Comparator): Internal osteogenesis distractor in acquired mandibular deformities in patients in growing age
  Interventions: Device: Internal Osteogenesis distractor
- II-A External distraction (Active Comparator): External osteogenesis distractor in acquired mandibular deformities in patients in growing age
  Interventions: Device: External Osteogenesis distractor
- II-B Internal distraction (Active Comparator): Internal osteogenesis distractor in acquired mandibular deformities in Adult patients.
  Interventions: Device: Internal Osteogenesis distractor
- II-B External distraction (Active Comparator): External osteogenesis distractor in acquired mandibular deformities in Adult patients.
  Interventions: Device: External Osteogenesis distractor

INTERVENTIONS:
Device: Internal Osteogenesis distractor — Internal distraction osteogenesis in mandible
  Arms: I-A Internal distraction; I-B Internal distraction; II-A Internal distraction; II-B Internal distraction
Device: External Osteogenesis distractor — External distraction osteogenesis in mandible
  Arms: I-A External distraction; I-B External distraction; II-A External distraction; II-B External distraction

SUMMARY:
Distraction osteogenesis is a powerful technique for creating new bone during significant lengthening of the mandible without the need for bone grafting and associated donor site morbidity.

The idea of distraction osteogenesis was largely abandoned by many until the 1950s. Ilizarov minimized complications by performing a corticotomy with minimal disruption of the surrounding blood supply and using a system of tension ring fixators to control the distraction in multiple planes. Through a series of experimental studies and clinical applications, Ilizarov established the foundation of distraction osteogenesis and its role in orthopedic management.

Applications in craniofacial surgery were first seen in 1973, when Synder et al applied the approach to mandibular lengthening in a canine animal model. Almost another 20 years passed before McCarthy and colleagues published, in 1992, the first report of mandibular lengthening in 4 children with congenital mandibular deficiency, 3 with hemifacial microsomia, and 1 with Nager syndrome. Thereafter, its role rapidly expanded to the midface and nearly all classic approaches to craniofacial reconstruction.

In general, mandibular distraction can be performed in the ramus for ramus lengthening, in the mandibular angle for downward and forward advancement, or in the mandibular body. Ramus or gonial angle distraction are mainly used to treat facial asymmetries as in hemifacial macrosomia.

Severe mandibular retrognathia can be classified as congenital or acquired. Congenital abnormalities that are associated with severe mandibular retrognathia or micrognathia include craniofacial syndromes such as hemifacial microsomia, Pierre-Robin syndrome, Treacher-Collins syndrome, and Nager syndrome. Adult patients with craniofacial syndromes may have undergone previous surgery at an earlier age, but unfavorable postsurgical growth or skeletal relapse may have occurred.

Severe mandibular retrognathia also can develop following maxillofacial trauma and mandibular fractures, which may have occurred in an adult or as a child Condylar fractures occurring at an early age can result in subsequent bony and/or fibrous temporomandibular joint ankylosis and/or deficient mandibular growth, also adult patients with complications from previous mandibular tumor resection and reconstruction can also present with acquired severe mandibular retrognathia that may require distraction osteogenesis as well.

Despite the advantages of extra-oral distraction devices in the hands of clinicians (application for very small children, simplicity of attachment, ease of manipulation, bidirectional and multidirectional dis- traction), patients are apprehensive about wearing bulky external appliances because of the social inconvenience and the potential of permanent facial scars, these disadvantages and limitations were the primary force driving the evolution of mandibular lengthening and widening toward the development of intra-oral devices.

However nowadays both internal and external distractors are used in a variety of indications in these cases each of the two types of distractor devices has its own advantages and disadvantages.

Aim of the work:

The aim of this study is to compare external and internal distraction devices for mandibular lengthening in terms of bone lengthening, patient comfort, and complications.

DETAILED DESCRIPTION:
The study will be conducted on 30 patients who are suffering mandibular problems either congenital acquired or post tumor mandibular resection that requires lengthening of the mandible, attending the outpatient clinic of Plastic Surgery Department in Ain Shams University Hospital & Assiut University Hospital.

Preoperative assessment:

* Informed consent will be obtained from all patients before their inclusion in the study.
* Photographs will be taken for the patient in lateral, antro-posterior and oblique positions preoperative.
* Lateral cephalometric radiographs or computed tomography (CT) or cone beam CT scans will be done for each patient pre-operatively.
* The decision to perform internal or external device will be based on preoperative and intraoperative considerations, such as anatomical bony characteristics affecting the possibility to place internal devices and patient cooperation.

Principles of the operation:

* anaesthesia: general anesthesia.
* Intraoperative consideration of internal versus external distractor is decided depending on the availability of bone stock.
* Osteotomy will be done according to each case individually making sure that it suits the vector of distraction required for each case.
* The approach for the external devices will be intraoral between the mental nerve anteriorly and gonial area posteriorly on both sides of the mandible.
* The approach for internal devices will be intraoral. While preserving the mandibular branch of the facial nerve.
* After 3-5 days of latency period for callus organization, gradual lengthening of the mandible will be performed at a rate of 0.5 mm twice a day for a total of 1 mm per day until achieving desired length.

Postoperative management and assessment:

* The patient will take broad spectrum and anaerobic antibiotics, anti-edematous, analgesic in addition to supportive treatment.
* After 3-5 days of latency period for callus organization according to patient age and condition, gradual lengthening of the mandible was performed at a rate of 0.5 mm twice a day for a total of 1 mm per day until achieving desired length.
* Following distraction phase there will be consolidation phase that will not be less than 8 weeks.
* Removing of internal or external distractor device and start retention phase if required with assistance of orthodontic appliances to avoid relapse.
* The patients will be evaluated with lateral cephalograms and head CT to assess the changes and amount of new bone formation following distraction.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females with congenital retrognathia or micrognathia.
2. Males and females between one month and 50 years.
3. Patients with acquired mandibular deformities as post traumatic (temporomandibular ankyloses), asymmetries, post-surgical as after mandibular tumor resection and irradiation.

Exclusion Criteria:

1. Patients with systemic illness as cardiac diseases, or mental disorders & hepatic patients (generally debilitating diseases).

Ages: 1 Month to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of bone formation | 6 months

SECONDARY OUTCOMES:
Failure | 1 month, 3months, 6months
  Failure of distraction will be assessed by the amount of bone formed in mm and the target rate of bone lenghtening to be achieved... e.g.. if the target is to lengthen 20mm we consider failure if the bone lengthening is less than 20mm
Complications | 1 week
  infection will be assessed for discharge around the pins if fever is present after operation this will be considered as infection from surgery, post-operative scars wether the scar is depressed hypertrophic or keloid forming scar, loosening of the pins wehter they remained in place or otherwise they are loosened

CONTACTS AND LOCATIONS:
Overall Officials: Assem Kamel, MD, Principal Investigator — Assiut University; Osama Taha, MD, Study Chair — Assiut University; Awny Askalany, MD, Study Chair — Assiut University; Ehab Ragab, M.Sc, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rachmiel A, Levy M, Laufer D. Lengthening of the mandible by distraction osteogenesis: report of cases. J Oral Maxillofac Surg. 1995 Jul;53(7):838-46. doi: 10.1016/0278-2391(95)90346-1. No abstract available. PMID 7595803
- [Background] Kaban LB, Padwa BL, Mulliken JB. Surgical correction of mandibular hypoplasia in hemifacial microsomia: the case for treatment in early childhood. J Oral Maxillofac Surg. 1998 May;56(5):628-38. doi: 10.1016/s0278-2391(98)90465-7. No abstract available. PMID 9590345